CLINICAL TRIAL: NCT06279104
Title: A Comparative Study of the Treatment of Real-world Patients With Clear Cell Carcinoma of the Ovary
Status: Recruiting | Type: Observational
Sponsor: Tongji Hospital (Other)
Collaborators: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Henan Cancer Hospital (Other Government); Qilu Hospital of Shandong University (Other); Hubei Cancer Hospital (Other); Anhui Provincial Cancer Hospital (Other); Peking University Cancer Hospital & Institute (Other); Hunan Province Tumor Hospital (Other); First Affiliated Hospital of Suzhou Medical College (Other); Shandong Tumor Hospital (Other); Chongqing University Cancer Hospital (Other); First Affiliated Hospital of Zhongshan Medical University (Other); Peking University Shenzhen Hospital (Other)
Responsible Party: Principal Investigator, Qinglei Gao, Prof., Tongji Hospital
Other Study IDs: 2023-TJ-OCCC
Record Dates: First submitted 2024-02-15; First posted 2024-02-26 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Ovarian Clear Cell Carcinoma
Keywords: Ovarian clear cell carcinoma; real world study; immune checkpoint inhibitor

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- real-world study (RWS)-Chemotherapy
  Interventions: Drug: physician's choice of chemotherapy
- RWS-ICI
  Interventions: Drug: immune checkpoint inhibitor based therapy

INTERVENTIONS:
Drug: physician's choice of chemotherapy — physician's choice of chemotherapy for relapsed/refractory ovarian clear cell carcinoma
  Groups: real-world study (RWS)-Chemotherapy
Drug: immune checkpoint inhibitor based therapy — immune checkpoint inhibitor based therapy for relapsed/refractory ovarian clear cell carcinoma
  Groups: RWS-ICI

SUMMARY:
The goal of this observational study is to learn about the treatment effectiveness of physician's choice of chemotherapy and the immune checkpoint inhibitor (ICI)-based therapy in patients with relapsed/refractory ovarian clear cell carcinoma (OCCC), and compare the treatment response with the phase II, single-arm clinical trial INOVA to investigate the efficacy of combinational therapy of sintilimab plus bevacizumab. The main questions it aims to answer are:

* What is the efficacy of physician's choice of chemotherapy in relapsed/refractory OCCC patients in the real world?
* Is ICI-based therapy more effective than physician's choice of chemotherapy in real-world for relapsed/refractory OCCC patients?
* Dose the combinational regimens of sintilimab plus bevacizumab in Sintilimab Plus Bevacizumab in Recurrent/Persistent Ovarian Clear Cell Carcinoma (INOVA) trial more effective than physician's choice of chemotherapy?

Participants will be respectively retrieved and extracted de-identified, longitudinal electronic health records (EHR)-derived data.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients with age ≥ 18 years old and ≤ 75 years old.
2. There must be a histological diagnosis of ovarian clear cell carcinoma.
3. Patients with recurrent or persistent ovarian clear cell carcinoma must have at least one-line pretreated platinum-containing chemotherapy.
4. Eastern Cooperative Oncology Group (ECOG) performance status score ≤ 2.
5. Expected survival time ≥ 12 weeks.

Exclusion Criteria:

1.Histological evidence of non-ovarian clear cell carcinoma.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with relapsed/persistent OCCC were extracted de-identified, longitudinal electronic health records (EHR)-derived data from 12 tertiary hospitals in China since October 2008. Consecutive patients were enrolled with no restriction on treatment regimens.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
tumor response rate | through study completion, an average of 1 year
  The tumor responses to treatment were evaluated by an independent central investigator according to RECIST version 1.1

SECONDARY OUTCOMES:
progression-free survival (PFS) | through study completion, an average of 1 year
  the time from therapy initiation to the first documented progression or death from any cause, whichever occurred first
time to response (TTR) | through study completion, an average of 3 months
  the time from therapy initiation to the first documented complete response or partial response
duration of response (DOR) | through study completion, an average of 1 year
  the time from the first documented response to disease progression or death, whichever occurs first
disease control rate (DCR) | through study completion, an average of 1 year
  the proportion of patients with complete response, partial response, and stable disease

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data will be available (including data dictionaries). The individual participant data that underlie the results reported in this article after deidentification (text, tables, figures, and appendices) in particular will be shared
Supporting Information: Study Protocol, SAP, ICF, CSR
URL: http://nuwa.com